CLINICAL TRIAL: NCT03208621
Title: Evaluation of PET and Laparoscopy in STagIng Advanced Gastric Cancer: a Multicenter Prospective Study
Brief Title: Evaluation of PET and Laparoscopy in STagIng Advanced Gastric Cancer
Acronym: PLASTIC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Nederlandse Vereniging voor Heelkunde (Unknown); Federatie Medisch Specialisten (Unknown); Patientfederatie Nederland (Unknown); Zorgverzekeraars Nederland (Unknown)
Responsible Party: Principal Investigator, Jelle P. Ruurda, Doctor, UMC Utrecht
Other Study IDs: 16-1633/C
Record Dates: First submitted 2017-06-30; First posted 2017-07-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Gastric Cancer; Staging; FDG-PET/CT; Diagnostic Laparoscopy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational group: The diagnostic tests to be investigated in this study is the use of PET and DLS in addition to the initial staging with gastroscopy and CT of patients with an advanced tumor (cT3-4)

SUMMARY:
Objective: To evaluate the impact and cost-effectiveness of FDG-PET/CT (PET) and diagnostic laparoscopy (DLS) in addition to initial staging by CT and gastroscopy in patients with advanced gastric cancer.

Hypothesis: The study hypothesizes that performing DLS and PET for advanced gastric adenocarcinomas results in a reduction in the number of futile gastrectomies performed and a favorable cost-effectiveness. According to the literature, in 27% of patients a futile gastrectomy can be prevented, and the annual cost-reduction is an estimated €916.438.

Study design: The study design is a prospective observational study. Study population: The study population consists of patients with a surgically resectable, advanced gastric adenocarcinoma (cT3-4a,N0-3,M0), that are scheduled for treatment with curative intent after initial staging with gastroscopy and CT.

Usual care / comparison: Both PET and DLS were recently included in the new Dutch guidelines for the treatment of gastric cancer, as staging modalities for advanced (T3-4) tumors after initial staging. The costs of the study population will be compared to retrospective data of patients who underwent curative surgery (gastrectomy) after initial staging with CT alone.

Outcome measures: The primary outcome of this study will be the proportion of patients in whom the PET or DLS lead to a change in treatment strategy. The accuracy of each modality will be analyzed separately. Secondary outcome parameters will be diagnostic performance, morbidity and mortality, quality of life, cost-reduction and cost-effectiveness.

Sample size: Based on the expectation that 22% of patients will have a change in treatment strategy, at least 239 patients will be needed for this study to demonstrate that the diagnostic modalities in the new guideline are break-even. Approximately 543 patients will be eligible for the study in 36 months.

Cost-effectiveness analysis: A state-of-the-art cost-effectiveness analysis and budget impact analysis will be performed on the additive value of PET and DLS by both prospective and retrospective data collection

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the stomach or esophagogastric junction (Siewert II and III), by gastroscopy.
* Underwent evaluation with computed tomography (CT) of the abdomen and chest.
* Surgically resectable, advanced tumor (cT3-4a,N0-3,M0), as determined by a multidisciplinary team meeting. An advanced tumor is defined as a transmural tumor with an irregular outer margin, objectified on CT.
* Intention to perform a curative gastrectomy

Exclusion Criteria:

* Siewert type I esophagogastric junction tumor
* Unfit or unwilling to undergo surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of patients with a surgically resectable, advanced gastric adenocarcinoma (cT3-4a,N0-3,M0), that are scheduled for treatment with curative intent after initial staging with gastroscopy and CT.
Sampling Method: Non-Probability Sample
Enrollment: 394 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in treatment strategy | 6 months after performing staging
  The primary outcome of this study will be the proportion of patients in whom the PET or DLS lead to a change in treatment strategy.

SECONDARY OUTCOMES:
Diagnostic performance | 6 months after performing staging
  Sensitivity, specificity, positive predictive value and negative predictive value of FDG/PET-CT and Diagnostic Laparoscopy
Morbidity | 3 months after performing staging
  Complications of staging modalities
Quality of life | Up to 5 years postoperative
  Quality of life with EORTC questionnaires
Cost-reduction | 12 months after performing staging
  Annual reduction in costs in the Netherlands of FDG-PET/CT and diagnostic laparoscopy, measured by reviewing hospital financial files and comparing with the previous situation without the staging
Cost-effectiveness | 12 months after performing staging
  Cost-effectiveness of FDG-PET/CT and diagnostic laparoscopy, measured by reviewing hospital financial files and comparing with the previous situation without the staging modalities
Mortality | 3 months after performing staging
  90-day mortality of the staging modalities

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smyth E, Schoder H, Strong VE, Capanu M, Kelsen DP, Coit DG, Shah MA. A prospective evaluation of the utility of 2-deoxy-2-[(18) F]fluoro-D-glucose positron emission tomography and computed tomography in staging locally advanced gastric cancer. Cancer. 2012 Nov 15;118(22):5481-8. doi: 10.1002/cncr.27550. Epub 2012 May 1. PMID 22549558
- [Derived] de Jongh C, van der Meulen MP, Gertsen EC, Brenkman HJF, van Sandick JW, van Berge Henegouwen MI, Gisbertz SS, Luyer MDP, Nieuwenhuijzen GAP, van Lanschot JJB, Lagarde SM, Wijnhoven BPL, de Steur WO, Hartgrink HH, Stoot JHMB, Hulsewe KWE, Spillenaar Bilgen EJ, van Det MJ, Kouwenhoven EA, Daams F, van der Peet DL, van Grieken NCT, Heisterkamp J, van Etten B, van den Berg JW, Pierie JP, Eker HH, Thijssen AY, Belt EJT, van Duijvendijk P, Wassenaar E, Wevers KP, Hol L, Wessels FJ, Haj Mohammad N, Frederix GWJ, van Hillegersberg R, Siersema PD, Vegt E, Ruurda JP; PLASTIC Study Group. Impact of 18FFDG-PET/CT and Laparoscopy in Staging of Locally Advanced Gastric Cancer: A Cost Analysis in the Prospective Multicenter PLASTIC-Study. Ann Surg Oncol. 2024 Jun;31(6):4005-4017. doi: 10.1245/s10434-024-15103-4. Epub 2024 Mar 25. PMID 38526832
- [Derived] Brenkman HJF, Gertsen EC, Vegt E, van Hillegersberg R, van Berge Henegouwen MI, Gisbertz SS, Luyer MDP, Nieuwenhuijzen GAP, van Lanschot JJB, Lagarde SM, de Steur WO, Hartgrink HH, Stoot JHMB, Hulsewe KWE, Spillenaar Bilgen EJ, van Det MJ, Kouwenhoven EA, van der Peet DL, Daams F, van Sandick JW, van Grieken NCT, Heisterkamp J, van Etten B, Haveman JW, Pierie JP, Jonker F, Thijssen AY, Belt EJT, van Duijvendijk P, Wassenaar E, van Laarhoven HWM, Wessels FJ, Haj Mohammad N, van Stel HF, Frederix GWJ, Siersema PD, Ruurda JP; PLASTIC Study Group. Evaluation of PET and laparoscopy in STagIng advanced gastric cancer: a multicenter prospective study (PLASTIC-study). BMC Cancer. 2018 Apr 20;18(1):450. doi: 10.1186/s12885-018-4367-9. PMID 29678145